CLINICAL TRIAL: NCT02794792
Title: A Phase 3, Double-blind, Randomized Study to Assess the Efficacy and Safety of Ipragliflozin in Combination With Metformin Compared to Metformin Plus Placebo in Subjects in Russia With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin
Brief Title: A Study to Assess the Efficacy and Safety of Ipragliflozin in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin
Acronym: IMPRESSION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1941-CL-9001
Record Dates: First submitted 2016-03-14; First posted 2016-06-09 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; ASP1941; Ipragliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metformin and placebo (Active Comparator): Participants will receive daily dosage of Metformin and Placebo as single tablets.
  Interventions: Drug: Metformin; Drug: Placebo
- Metformin and Ipragliflozin (Experimental): Participants will receive daily dosage of Metformin and Ipragliflozin (2 dose strengths) as single tablets.
  Interventions: Drug: Ipragliflozin L-proline; Drug: Metformin
- Metformin, placebo and Ipragliflozin (Other): Participants will receive daily dosage of Metformin, placebo and Ipragliflozin (1 dose strength) as single tablets.
  Interventions: Drug: Ipragliflozin L-proline; Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Ipragliflozin L-proline — Oral
  Other Names: Suglat; ASP1941
  Arms: Metformin and Ipragliflozin; Metformin, placebo and Ipragliflozin
Drug: Metformin — Oral
  Other Names: Riomet; Glucophage; Glumetza; Glucophage XR; Fortamet
Drug: Placebo — Oral
  Arms: Metformin and placebo; Metformin, placebo and Ipragliflozin

SUMMARY:
The main purpose of this study is to evaluate the efficacy in reducing glycated hemoglobin of ipragliflozin in combination with metformin compared with metformin plus placebo in subjects with type 2 diabetes mellitus who have inadequate glycemic control on metformin.

DETAILED DESCRIPTION:
This is a phase 3, double-blind, randomized study to assess the efficacy and safety of ipragliflozin in combination with metformin compared to metformin plus placebo in subjects in Russia with type 2 diabetes mellitus who have inadequate glycemic control on metformin. Subjects will enter a 10-day (± 3 days) screening period, followed by a 2-week single-blind placebo run-in period, followed by a 24-week randomized double-blind treatment period and a 4-week follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with type 2 diabetes mellitus at least 12 weeks before visit 1.
* Subject has been on a stable dose and a daily dose regimen of metformin ≥ 1500 mg for at least 12 weeks prior to visit 1.
* Subject has HbA1c ≥ 7.5% and ≤ 11.0% at visit 1.
* Subject has been on a stable diet and exercise program for at least 12 weeks prior to visit 1 and is willing to maintain this program for the duration of the treatment period.
* Subject has a body mass index (BMI) of 20 to 45 kg/m2, inclusive, at visit 1.
* Subjects are allowed to continue taking their medication for concomitant diseases (including over-the-counter products), provided they have been on a stable dose for a minimum of 30 days prior to visit 1.
* Female subjects must either:

  1. Be of non-childbearing potential:

     * postmenopausal (defined as at least 1 year without any menses) prior to screening, or
     * documented as surgically sterile
  2. Or, if of childbearing potential,

     * Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
     * And have a negative serum pregnancy test at visit 1
     * And, if heterosexually active, agree to consistently use 2 forms of highly effective birth control (at least 1 of which must be a barrier method) starting at screening, throughout the study period and for 28 days after the final study drug administration.
* Female subjects must agree not to breastfeed starting at screening, throughout the study period and for 28 days after the final study drug administration.
* Female subjects must not donate ova starting at screening, throughout the study period and for 28 days after the final study drug administration.
* Male subjects and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (at least 1 of which must be a barrier method) starting at screening and continue throughout the study period.
* Male subjects must not donate sperm starting at screening and throughout the study period.

Exclusion Criteria:

* Subject has type 1 diabetes mellitus.
* Subject has received any medication for glycemic control, with the exception of metformin, (e.g., oral antidiabetic drugs, insulin, etc.) within 12 weeks prior to visit 1.
* Subject is currently receiving an excluded medication or has received insulin within 12 weeks prior to visit 1 or during the screening period.
* Subject has a history of stroke, unstable angina, myocardial infarction, any vascular intervention or heart failure (New York Heart Association Class III-IV;) within 12 weeks prior to visit 1.
* Subject has had a malignancy in the last 5 years, except for adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Subject has a history of diabetic coma or precoma.
* Subject has a history of ketoacidosis or lactic acidosis.
* History of drinking more than 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) (> 14 units of alcohol for female subjects) or history of drugs abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates) within 3 months prior to visit 1.
* Subject is known to have hepatitis or be a carrier of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or is known to be positive for human immunodeficiency virus (HIV)-1 and/or HIV-2.
* Subject has a severe infection, has serious trauma, or is a perioperative subject.
* Subject has symptomatic urinary tract infection or genital infection at visit 1 and/or just prior to randomization at visit 3.
* Subject has uncontrolled severe hypertension (or subject whose systolic blood pressure is > 180 mmHg or diastolic blood pressure of > 110 mmHg measured in a sitting position after 5 minutes of rest at visit 1).
* Subject has an alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2 x the upper limit of normal (ULN) range or has a total bilirubin > 1.5 x ULN at visit 1.
* Subject has a urinary microalbumin/creatinine ratio ≥ 300 mg/g at visit 1.
* Subject has estimated glomerular filtration rate (GFR) value of < 60 mL/min/1.73 m2 at visit 1 (using the Modification of Diet in Renal Disease [MDRD] calculation).
* Subject has known or suspected hypersensitivity to ipragliflozin or any components of the formulations used or a history of allergy for Sodium-glucose cotransporter (SGLT)2 inhibitors.
* Subject has previously received ipragliflozin or other SGLT2 inhibitors.
* Subject is concurrently participating in another drug study or has received an investigational drug within 30 days or the limit set by national law, whichever is longer, prior to visit 1 or plans to receive another investigational drug during the study.
* Female subject who is currently pregnant or lactating
* Male or female subject who does not use appropriate contraception during the study.
* The subject is unable to adhere to the treatment regimen, protocol procedures or study requirements (including discontinuation criteria during the run-in period), in the investigator's judgment.
* Subject has an unstable medical or psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c with ipragliflozin once daily added on to metformin compared to placebo added on to metformin | Baseline and 12 weeks
  Glycated hemoglobin (HbA1c)

SECONDARY OUTCOMES:
Change from baseline in HbA1c in each treatment group | Baseline and 24 weeks
Change from baseline in FPG in each treatment group | Baseline, 12 weeks and 24 weeks
  Fasting plasma glucose (FPG)
Number of patients reaching a treatment goal in HbA1c of < 7.0% in each treatment group | Up to 24 weeks
Change in body weight in each treatment group | Baseline, 12 weeks and 24 weeks
Change in blood pressure in each treatment group | Baseline, 12 weeks and 24 weeks
Number of patients with AEs | Up to 24 weeks
  Adverse Events (AEs)
Number of patients with AEs of special interest | Up to 24 weeks
  AEs of special interest include: hypoglycemic events, dehydration/hypovolemia, urinary tract infections and genital infections
Percentage of patients reaching a treatment goal in HbA1c of < 7.0% in each treatment group | Up to 24 weeks
Change from baseline in PROs as measured by European Quality of Life 5 Dimensions 5 Levels [EQ-5D-5L] questionnaire | Baseline, 12 weeks and 24 weeks
  Patient-reported outcomes (PROs)
Change from baseline in PROs as measured by Audit of Diabetes Dependent Quality of Life [ADDQoL-19] questionnaire | Baseline, 12 weeks and 24 weeks
Change from baseline in PROs as measured by Work Productivity and Activity Impairment: General Health [WPAI:GH] questionnaire | Baseline, 12 weeks and 24 weeks
Change from baseline in PROs as measured by Diabetes Medication Satisfaction [Diab-MedSat] questionnaire | Baseline, 12 weeks and 24 weeks
Percentage of patients with AEs | Up to 24 weeks
Percentage of patients with AEs of special interest | Up to 24 weeks
  AEs of special interest include: hypoglycemic events, dehydration/hypovolemia, urinary tract infections and genital infections

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Europe B.V.
Locations (14):
- Russia (14):
  - Site RU70011, Moscow
  - Site RU70005, Moscow
  - Site RU70003, Moscow
  - Site RU70009, Moscow
  - Site RU70010, Nizhny Novgorod
  - Site RU70008, Saint Petersburg
  - Site RU70014, Saint Petersburg
  - Site RU70007, Saint Petersburg
  - Site RU70002, Saint Petersburg
  - Site RU70006, Samara
  - Site RU70004, Saratov
  - Site RU70015, Volgograd
  - Site RU70001, Yaroslavl
  - Site RU70013, Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=255